CLINICAL TRIAL: NCT03870282
Title: Increasing Childhood Sleep Duration in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 18-015830
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sleep
Keywords: Childhood sleep promotion; Sleep promotion; Sleep

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- 9h 15m Goal (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive B | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive B | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive B | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A&B | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentive A&B | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- 9h 15m Goal | Incentives A&B | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive B | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive B | Text A (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive B | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A&B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A&B | Texts B (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentive A&B | Texts A (Experimental)
  Interventions: Behavioral: Sleep Extension
- Personal Goal | Incentives A&B | Texts A&B (Experimental)
  Interventions: Behavioral: Sleep Extension

INTERVENTIONS:
Behavioral: Sleep Extension — The intervention is designed to test if sleep tips delivered by text messages can aid with reaching sleep targets. And if additional motivational text messages can further aide with reaching sleep targets.

SUMMARY:
Investigators seek to determine if a mobile health based intervention can be developed to target increases in childhood sleep duration.

DETAILED DESCRIPTION:
Investigators seek to determine if an online based intervention can be developed to target increases in childhood sleep. The primary objectives of this study are to determine if different messaging strategies lead to the longer sleep duration.Children aged 9-12 who sleep about 6-8.5 hours per night will wear a Fitbit for 11 weeks in order to measure sleep patterns. Participants will have a sleep goal to meet each night. Participants will be randomized to one of thirty-two study conditions and receive text and/or email messaging. Some study arms receive additional messaging with different content and frequency of delivery. The study involves one visit to the Children's Hospital of Philadelphia (CHOP).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 9 to 12 years.
2. Speak, read and write in English.
3. Parental/guardian permission (informed consent) and child assent.
4. Have a computer or a tablet computer with access to the Internet, or own a smartphone with a data and text plan.
5. Parent reported time in bed on school nights between 6.0-8.5 hours in bed at night (e.g. 7-hour time in bed: go to bed at 11pm & get out of bed at 6am).

Exclusion Criteria:

1. Any clinically diagnosed sleep disorder (e.g. sleep apnea).
2. Diagnosed with a psychiatric disorder [e.g. attention deficit hyperactivity disorder (ADHD), depression, anxiety].
3. Diagnosed with an eating disorder.
4. Musculoskeletal or neurological disorder that limits physical movement and activity.
5. Use of medications (prescription or otherwise) known to affect body weight and/or sleep.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Actigraphy Estimated Weeknight Sleep Duration | 10 weeks
  The investigators' primary outcome is actigraphy estimated weeknight sleep duration operationalized as the average hours per weeknight per week.

SECONDARY OUTCOMES:
Sleep Disturbance Score | 15 minutes
  Measured using the validated Patient-Reported Outcomes Measurement Information System (PROMIS) 9-item bank for pediatric sleep, ages 8-17y. The sleep disturbance score is calculated by summing responses to items related to sleep onset, sleep continuity and sleep quality. Higher scores for sleep disturbance indicate poorer sleep quality. We will operationalize our secondary outcomes as T-scores, using the standard PROMIS approach.
Sleep Related Impairment Score | 15 minutes
  Measured using the validated Patient-Reported Outcomes Measurement Information System (PROMIS) 9-item bank for pediatric sleep, ages 8-17y. The sleep-related impairment score is calculated by summing responses to items related to daytime sleepiness, cognition, affect & behavior and daytime activities. Higher scores for sleep impairment indicate poorer sleep quality. We will operationalize our secondary outcomes as T-scores, using the standard PROMIS approach.

OTHER OUTCOMES:
Actigraphy Estimated Nighttime Sleep Duration | 10 weeks
  The investigators' other outcomes are actigraphy estimated nighttime sleep duration operationalized as the average hours per night per week.
Actigraphy Estimated Weekend Night Sleep Duration | 10 weeks
  The investigators' other outcomes are actigraphy estimated weekend night sleep duration operationalized as the average hours per weekend night per week.
Actigraphy Estimated Sleep Efficiency (Nighttime, Weeknight and Weekend Night) | 10 weeks
  The investigators' other outcomes are actigraphy estimated sleep efficiency per night, weeknight, and weekend night operationalized as percentage of time spent asleep during the overnight sleep period.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Mitchell, PhD, Principal Investigator — Childern's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No